CLINICAL TRIAL: NCT01383889
Title: Acute Effects on the Mother and Fetus in Two Modalities of Exercise in Pregnancy: a Randomized Controlled Trial.
Brief Title: Acute Maternal and Fetal Effects of Exercise in Pregnancy
Acronym: EXPREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Collaborators: Professor Fernando Figueira Integral Medicine Institute (Other); Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Isabela Coutinho, Professor, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: EXPREG 2011
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Blood Pressure; Heart Rate and Rhythm Disorders; Hypoglycemia; Lactate; Nitrate; Cholesterol (Total and HDL); Abnormality in Fetal Heart Rate or Rhythm, Unspecified as to Episode of Care
Keywords: Physical exercise; Pregnancy; Fetal well being
MeSH Terms: conditions — Hypoglycemia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treading mill exercise (Other): Pregnant women in this group will perform treadmill exercise during 20 minutes. The intensity of exercise will be maintained between 60% and 80% of maximum heart rate by Karvonen formula, in addition to the subjective perception of exertion on the modified Borg scale (moderate intensity).
  Interventions: Other: Physical exercise
- Stationary bicycle exercise (Other): Pregnant women in this group will perform exercise using a stationary bicycle. The intensity of exercise will be maintained between 60% and 80% of maximum heart rate by Karvonen formula, in addition to the subjective perception of exertion on the modified Borg scale (moderate intensity).
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Two modalities of exercise will be compared: treading mill and stationary bicycle. Pregnant women enrolled in the study will perform exercise during 20 minutes and will be monitored 20 minutes before, during and 20 minutes after exercise.

SUMMARY:
This will be an open randomized clinical trial involving pregnant women between 35 and 37 weeks randomized to two modalities of exercise: treadmill or stationary bike. The study hypothesis is that exercise on a stationary cycle causes less maternal and fetal effects in relation to treadmill exercise.We will study the acute effects of exercise for both the mother and the fetus, monitoring the parameters before, during and after exercise for 20 minutes. The exercise intensity will be moderate, remaining between 60% and 80% of maximum heart rate. Women will be monitored with a recording equipment of ABPM (ambulatory blood pressure monitorization) and continuous cardiotocography and blood will be collected to measure blood glucose, total cholesterol and HDL, nitrate and lactate before, during and after exercise. The analysis variables are: maternal heart rate and blood pressure, fetal heart rate, number of fetal movements, transient accelerations, decelerations, short-term variability, episodes of high variability, uterine tone, glucose, lactate, nitrate, total cholesterol and HDL.The analysis will be based on intention to treat, according to the recommendations of the CONSORT (2010).

DETAILED DESCRIPTION:
Background: Exercise has been encouraged during pregnancy in order to reduce undesirable outcomes such as pre-eclampsia, excessive weight gain and diabetes. Despite widespread among pregnant women and obstetricians, little is known about the acute effects for both mother and fetus at the time of exercise, with most existing research controlling only the pre-and post-exercise.

Objective: To study the acute effects of two moderate modalities of exercise on the pregnant woman and fetus.

Methods: This will be an open randomized controlled trial to be conducted in Campina Grande, Brazil, from December 2011 to December 2012. The pregnant women with gestational age between 35 and 37 weeks will be randomized into two groups of moderate-intensity exercise: treadmill and stationary bicycle. Pregnant women and fetuses will be monitored for 60 minutes divided in three steps of 20 minutes each: baseline assessment, monitoring during exercise and recovery period. Women will be monitored using a recording equipment of ABPM (ambulatory blood pressure monitorization) and fetal heart rate will be monitored through computerized cardiotocography. Blood will be collected to measure blood glucose, total cholesterol and HDL, nitrate and lactate before, during and after exercise. The intensity of exercise will be maintained between 60% and 80% of maximum heart rate by Karvonen formula, in addition to the subjective perception of exertion on the modified Borg scale (moderate intensity). During the monitoring period (in the three moments mentioned above) blood will be collected for the measurement of glucose, total cholesterol and HDL, nitrate and lactate. The analysis variables are: maternal heart rate and blood pressure, fetal heart rate, number of fetal movements, transient accelerations, decelerations, short-term variability, episodes of high variability, uterine tone, glucose, lactate, nitrate, total cholesterol and HDL

Statistical Analysis: Statistical analysis will be performed using Epi Info 3.5.3 and Medcalc 11.6.6.0 or higher versions available at the time. The analysis will be based on intention to treat, according to the recommendations of the CONSORT (2010). For comparison of levels of glucose, lactate, cholesterol, nitrate, maternal blood pressure, maternal and fetal heart rate, fetal movements, transient accelerations, decelerations, changes in short-term episodes of high variation, and uterine tone in the two groups a parametric test will be used (Student's t) if these variables have normal distribution, otherwise they will be evaluated using the nonparametric test of Mann-Whitney. To determine the association between mode of exercise and frequency of fetal bradycardia the chi-square test of association (Pearson) will be used at a 5% significance level. The risk ratio (RR) will be calculated as a measure of relative risk, as well as its 95% confidence interval. If a significant difference in the rate of bradycardia will be demonstrated between the groups, the NNH (Number Need Harm) will be calculated.

Ethical issues: The research project was approved by Institutional Review Board under the number CAAE 0195.0.133.000-11 All the participants will be informed about the objectives of the research and only will be included if they agree voluntarily to participate and sign an informed consent term. There are no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* Alive fetus
* Gestational age between 35 and 37 weeks
* Previous sedentarity

Exclusion Criteria:

* Smoking
* Chronic maternal illness
* Diseases that affect respiratory capacity
* Physical handicap precluding performing exercise
* Arterial Hypertension
* Diabetes in Pregnancy
* Placenta praevia
* Preterm labor
* Bleeding in the third trimester
* Fetal Growth Restriction
* Oligo-hydramnios
* Brain-sparing effect
* Fetal malformations
* Medical contraindications for performing exercise

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fetal bradycardia | 60 minutes
  Fetal heart rate will be monitored durante 60 minutes, 20 minutes before, 20 minutes during and 20 minutes after two modalities of exercise: treading mill and stationary bicycle. The frequency of fetal bradycardia will be assessed.

SECONDARY OUTCOMES:
Maternal blood pressure | 60 minutes
  Maternal blood pressure will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise)
Maternal heart rate | 60 minutes
  Maternal heart rate will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise)
Glycemia | 60 minutes
  Maternal glycemia will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise)
Maternal lactate | 60 minutes
  Maternal heart rate will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise)
Maternal nitrate | 60 minutes
  Maternal nitrate will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise)
Total Cholesterol and HDL | 60 minutes
  Total Cholesterol and HDL will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise)
Fetal heart rate | 60 minutes
  Fetal heart rate will be monitored during 60 minutes (20 minutes before, 20 minutes during and 20 minutes after the exercise). The following parameters will be assessed: fetal heart rate, bradycardia, fetal movements, transient accelerations, decelerations, changes in short-term episodes of high variation
Uterine tone | 60 minutes
  Uterine tone will be assessed 20 minutes before, 20 minutes during and 20 minutes after exercise

CONTACTS AND LOCATIONS:
Overall Officials: Melania MR Amorim, MD, PhD, Principal Investigator — Instituto Materno Infantil Prof. Fernando Figueira
Locations (1):
- Instituto Paraibano de Pesquisa Prof. Joaquim Amorim Neto, Campina Grande, Paraíba, Brazil